CLINICAL TRIAL: NCT07042308
Title: Natural History of Advanced Chronic Liver Diseases and Factors Associated With Hepatic Events - a Registry Study
Brief Title: Natural History of Advanced Chronic Liver Diseases
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Jimmy Che-To Lai, Assistant Professor (Clinical), Chinese University of Hong Kong
Other Study IDs: 2024.258
Record Dates: First submitted 2025-06-17; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Cirrhosis; Advanced Chronic Liver Disease
Keywords: advanced chronic liver disease
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Store 10 mL of clotted blood and 10 mL of EDTA blood for exploration or novel biomarkers, future genetic and biochemical research
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with advanced chronic liver disease: Adult patients with advanced chronic liver disease
  Interventions: Diagnostic Test: Transient elastography

INTERVENTIONS:
Diagnostic Test: Transient elastography — Liver stiffness and spleen stiffness from transient elastography

SUMMARY:
This is a retrospective-prospective registry cohort study. Patients with advanced chronic liver disease (ACLD) will be prospectively invited to this study. The study follow-up duration will be 10 years. The primary outcome is incident hepatic events and liver-related mortality. Participants will undergo annual transient elastography examination.

DETAILED DESCRIPTION:
Chronic liver diseases (CLD) has burdened the global healthcare system throughout the years. Among all causes of CLD, chronic hepatitis B (CHB) is generally the commonest cause of CLD in the Asia-Pacific region but the prevalence is expected to decline due to effective antiviral treatment. Similarly, with the introduction of direct-acting antiviral (DAA), chronic hepatitis C (CHC) is now readily curable. On the other hand, an increasing trend is observed in metabolic dysfunction-associated steatotic liver disease (MASLD) and alcohol-related liver disease (ARLD) which is likely to change the landscape of CLD both in the region and worldwide.

Advanced chronic liver disease (ACLD) or cirrhosis is a final common pathway of all CLD and was the 9th and 15th leading cause of death in Southeast Asia (0.42 million deaths) in 2019 as reported by the World Health Organization (WHO) Global Health Estimates. It also significantly increases the risk of hepatocellular carcinoma (HCC). With its significant impact on morbidity and mortality, the prognosis of compensated and decompensated states differ drastically and the field is pushing forward ways to prevent hepatic decompensation in order to improve liver-related outcomes. Non-selective beta-blockers (NSBB) has been shown to reduce risk of hepatic decompensation in patients with compensated advanced chronic liver disease (cACLD) and concomitant clinically significant portal hypertension (CSPH). Some other drugs including angiotensin converting enzyme inhibitor (ACEI)/angiotensin-receptor blocker (ARB), statin etc. have been shown in retrospective studies to reduce risk of hepatic decompensation but more evidence is required to draw conclusive interpretation.

Apart from medications, non-invasive tests (NIT), including liver stiffness measurement (LSM) and spleen stiffness measurement (SSM) from vibration-controlled transient elastography (VCTE) help prognosticate chronic liver diseases. Yet more validation is required on certain conditions such as in patients with obesity as well as HCC. Biomarkers are also under the spotlights for risk prediction but are yet to reach the stage for widespread clinical practice. Hence these areas deserve further studies.

Hong Kong is an area endemic for chronic hepatitis B as well as expected for an increase with MASLD and ARLD. There has not been an established registry to capture these ACLD patients for systematic monitoring and analysis. Thus, a registry for ACLD is imperative.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or above
* Known ACLD, defined by:

  * LSM > 10kPa or
  * Clinical cirrhosis, suggested by 1. ultrasonography of the hepatobiliary system shows features of cirrhosis (e.g. shrunken and nodular liver) and portal hypertension (e.g. dilated portal vein, portal-systemic collaterals or varices, splenomegaly, ascites). 2. Oesophagogastroduodenoscopy (OGD) shows presence of oesophageal varices (OV) and/or gastric varices (GV) and/or portal hypertensive gastropathy.

Exclusion Criteria:

* Current or past history of hepatocellular carcinoma (HCC)
* History of liver transplantation
* Asplenism or history of splenectomy
* Serious medical illness with limited life expectancy of less than 6 months
* Pregnancy
* Unable to obtain or refusal of informed consent from patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The prospective cohort will comprise of consecutive patients with advanced chronic liver disease attending hepatology clinics or in-patient care in Prince of Wales Hospital in Hong Kong. All patients will be screened if the eligibility criteria are fulfilled.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2035-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Incident hepatic events and liver-related mortality | 10 years
  Incident hepatic events (including ascites, variceal bleeding and overt hepatic encephalopathy) and liver-related mortality

SECONDARY OUTCOMES:
Incidence rate of each hepatic event | 10 years
  Hepatic events include ascites, variceal bleeding and overt hepatic encephalopathy
Incidence rate of hepatocellular carcinoma | 10 years
  Development of hepatocellular carcinoma
Changes in Child-Pugh and Model for End-stage Liver Disease scores | 10 years
  The minimum and maximum Child-Pugh score are 5 and 15, respectively. The minimum and maximum Model for End-stage Liver Disease score are 6 and 40, respectively. A higher score denotes worse outcome in both scores
Change in liver and spleen stiffness | 10 years
  Change in liver and spleen stiffness by transient elastography
Exploratory outcome on identification of novel biomarkers | 10 years
  Novel biomarkers include multi-omics exploration in relation to the primary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jimmy CT Lai, MB ChB, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Data may be shared upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months after the first publication until 15 years after the end of the study
Access Criteria: By email communication.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-23): https://cdn.clinicaltrials.gov/large-docs/08/NCT07042308/Prot_SAP_000.pdf
  • Informed Consent Form (2024-05-23): https://cdn.clinicaltrials.gov/large-docs/08/NCT07042308/ICF_001.pdf